CLINICAL TRIAL: NCT02306187
Title: The Effectiveness of Eldecalcitol in the Osteoporotic Patients Who Are Bisphosphonate Non-responders After Long-term Bisphosphonate Treatment
Brief Title: The Effectiveness of Eldecalcitol in the Bisphosphonate Non-respondered-patients With Osteoporosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Assistant Professor, Shinshu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BP-ED study 2014
Record Dates: First submitted 2014-11-24; First posted 2014-12-03 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
Keywords: The changes of bone mineral density and bone turnover markers
MeSH Terms: conditions — Osteoporosis | interventions — eldecalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Alfacaocidol (Experimental): Ahead of Eldecalcitol treatment, this group has not taken Alfacaocidol before. Eldecalcitol: the commercial name is Edirol We prescribe Edirol 0.5 or 0.75ug per day into each patient.
  Interventions: Drug: Edirol
- Alfacalcidol (Experimental): Ahead of Eldecalcitol treatment, this group has taken Alfacaocidol before. Eldecalcitol: the commercial name is Edirol We prescribe Edirol 0.5 or 0.75ug per day into each patient.
  Interventions: Drug: Edirol

INTERVENTIONS:
Drug: Edirol — Edirol 0.5 or 0.75ug once every day oral treatment for at least 1 year after initial visit.
  Other Names: Eldecalcitol

SUMMARY:
In the patients with osteoporosis, bisphosphonates (BPs) are a golden standard treatment. However, the bone turnover markers or the bone mineral density (BMD) are not improved in some osteoporotic patients even though they have taken BPs and alfacalcidol more than several years. In those case, the investigators better off prescribing BPs and Eldecalcitol, instead of BPs and Alfacalcitol.

DETAILED DESCRIPTION:
Alfacalcitol and Eldecalcitol are the similar vitamin D drugs. However, Eldecalcitol is an improved vitamin D drug than Alfacalcitol. Therefore, we investigate the effectiveness of Eldecalcitol in this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Osteoporosis
* Must be able to swallow tablets

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with bone turnover markers as a Measure of bone quality | At 4 months after the initial treatment
  Bone formation and bone absorption markers will be evaluated at each time point
Number of Participants with bone turnover markers as a Measure of bone quality | At 1 year after the initial treatment
  Bone formation and bone absorption markers will be evaluated at each time point

SECONDARY OUTCOMES:
Number of Participants with bone mineral density as a Measure of bone quality | At 4 months after the initial treatment
  Bone mineral density will be evaluated at each time point
Number of Participants with bone mineral density as a Measure of bone quality | At 1 year after the initial treatment
  Bone mineral density will be evaluated at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Yukio Nakamura, MD, PhD, Principal Investigator — Shinshu University School of Medicine
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan